CLINICAL TRIAL: NCT06088368
Title: Investigation of the Efficacy of Different Types of Lumbar Plexus Block Applied With Ultrasound-guided Shamrock Method
Brief Title: Lumbar Plexus Block Application in Ultrasound-guided Shamrock Method
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Bursa Yuksek Ihtisas Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Korgün Ökmen, Principal Investigator, Bursa Yuksek Ihtisas Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-3/7
Record Dates: First submitted 2023-10-12; First posted 2023-10-18 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Femoral Neck Fractures; Lumbosacral Plexus; Nerve Block
MeSH Terms: conditions — Femoral Neck Fractures

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- in-plane needle guidance (Active Comparator): Ultrasound -guided lumbar plexus block
  Interventions: Procedure: in-plane needle guidance
- out-of-plane needle guidance (Active Comparator): Ultrasound -guided lumbar plexus block
  Interventions: Procedure: out-of-plane needle guidance

INTERVENTIONS:
Procedure: in-plane needle guidance — Ultrasound -guided lumbar plexus block with in-plane needle guidance using the Shamrock method
  Arms: in-plane needle guidance
Procedure: out-of-plane needle guidance — Ultrasound -guided lumbar plexus block with out-of-plane needle guidance using Shamrock method
  Arms: out-of-plane needle guidance

SUMMARY:
The more effective use of ultrasound in regional anaesthesia techniques has made different block applications possible. Lumbar plexus block is also used for post-operative analgesia and surgical anaesthesia. Currently, in-plane ultrasound-guided LPB is widely used in short-axis imaging and Shamrock imaging.

DETAILED DESCRIPTION:
The purpose of this use is to investigate the effectiveness of lumbar plexus block application applied with in-plane and out-of-plane methods accompanied by Shamrock imaging.

ELIGIBILITY:
Inclusion Criteria:

* 18-90 years old
* ASA (American Society of Anaesthesiologist) Score I-III risk class
* Patients who will undergo femoral neck fracture operation.

Exclusion Criteria:

* Local Anaesthetic Allergy
* With Bleeding Diathesis Disorder
* Mental Disorders
* Allergic to the medicines used
* Previous Cerebrovascular Disease
* Body Mass Index above 30

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-10-20 (Estimated); Primary Completion 2024-01-25 (Estimated); Study Completion 2024-02-13 (Estimated)

PRIMARY OUTCOMES:
Block application time | up to 20 minutes
  The stopwatch will be started by another researcher with the needle skin penetration and the stopwatch will be stopped as soon as the needle leaves the skin.

SECONDARY OUTCOMES:
Number of interventions | up to 20 minutes
  intervention from the same or another site after exiting the skin
The number of needle guidance | up to 20 minutes
  Retraction and re-advancement of the needle after skin entry without exiting the skin
sensory block | up to 40 minutes
  Both lower limbs sensory block time after the applied block will be evaluated by pinprick and cold test (10.15., 20., 25., 30., 35. and 40 minutes).
motor block | up to 40 minutes
  Both lower limbs Modified Bromage scale was used to evaluate motor block. Modified Bromage scale 0 No motor block
  1. Raises the knee in flexion
  2. Raises the ankle
  3. Full block, can't move his foot

CONTACTS AND LOCATIONS:
Overall Officials: Korgün Ökmen, Assoc. PhD., Principal Investigator — Sağlık Bilimleri Üniversitesi Bursa Yüksek İhtisas Eğitim Ve Araştırma Hastanesi
Locations (1):
- University of Health Sciences,,Bursa Yuksek Ihtisas Training and Research Hospital,, Bursa, Turkey (Türkiye)